CLINICAL TRIAL: NCT01516580
Title: Intergroup Trial for Children or Adolescents With B-Cell Non Hodgkin Lymphoma or B-Acute Leukemia: Evaluation of Rituximab Efficacy and Safety in High Risk Patients - Phase III Trial
Brief Title: Intergroup Randomized Trial for Children or Adolescents With B-Cell Non Hodgkin Lymphoma or B-Acute Leukemia: Rituximab Evaluation in High Risk Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Inter B-NHL Ritux 2010 Phase 3; 2010-019224-31 (EudraCT Number)
Record Dates: First submitted 2012-01-19; First posted 2012-01-25 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: B-cell Non Hodgkin Lymphoma; Mature B-cell Leukemia Burkitt-type
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma | interventions — Vincristine; Cyclophosphamide; Methotrexate; Doxorubicin; Cytarabine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMB chemo (Active Comparator): Prephase (COP) for all groups followed by:
  * in group B: 4 courses: 2 COPADM + 2 CYM, with MTX 3g/m²
  * in group C: 6 courses: 2 COPADM + 2 CYVE + 2 maintenance courses, with MTX 8g/m², in 4h in C1, in 24h in C3 (except the 1st course) and CNS positive patients receive additional IT before each CYVE courses and HDMTX between CYVE courses.
  Interventions: Drug: Vincristine, cyclophosphamide, methotrexate, doxorubicin, cytarabine, ara-C
- LMB chemo + Rituximab (Experimental): LMB chemo as in the comparator arm Rituximab 375 mg/m² i.v.: 6 injections: two doses at 48h interval are given at D-2 and D1 of the 2 first courses (COPADM) and one dose at the beginning of the 2 following courses (CYM or CYVE).
  Interventions: Drug: Rituximab, Vincristine, cyclophosphamide, methotrexate, doxorubicin, cytarabine, ara-C

INTERVENTIONS:
Drug: Vincristine, cyclophosphamide, methotrexate, doxorubicin, cytarabine, ara-C — Prephase (COP) for all groups followed by:
  in group B: 4 courses: 2 COPADM + 2 CYM, with MTX 3g/m² in group C: 6 courses: 2 COPADM + 2 CYVE + 2 maintenance courses, with MTX 8g/m², in 4h in C1, in 24h in C3 (except the 1st course) and CNS positive patients receive additional IT before each CYVE courses and HDMTX between CYVE courses.
  Arms: LMB chemo
Drug: Rituximab, Vincristine, cyclophosphamide, methotrexate, doxorubicin, cytarabine, ara-C — LMB chemo as in the comparator arm Rituximab 375 mg/m² i.v.: 6 injections: two doses at 48h interval are given at D-2 and D1 of the 2 first courses (COPADM) and one dose at the beginning of the 2 following courses (CYM or CYVE).
  Arms: LMB chemo + Rituximab

SUMMARY:
The aim of the trial is to test whether adding 6 injections of rituximab to standard "Lymphome malin B" LMB chemotherapy regimen improves the Event Free Survival (EFS) compared with LMB chemotherapy alone in children / adolescents with advanced stage B-cell Non-Hodgkin Lymphoma (NHL) / B-Acute Leukemia (B-AL)(stage III and LDH > Nx2, any stage IV or B-AL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven B-cell malignancies, either Burkitt lymphoma or B-AL (=Burkitt leukaemia = L3-AL) or diffuse large B-cell NHL or aggressive mature B-cell NHL non other specified or specifiable.
* Stage III with elevated LDH level ("B-high"), [LDH > twice the institutional upper limit of the adult normal values (> Nx2)] or any stage IV or B-AL.
* 6 months to less than 18 years of age at the time of consent.
* Males and females of reproductive potential must agree to use an effective contraceptive method during the treatment, and after the end of treatment: during twelve months for women, taking into account the characteristics of rituximab and during five months for men, taking into account the characteristics of methotrexate.
* Complete initial work-up within 8 days prior to treatment that allows definite staging.
* Able to comply with scheduled follow-up and with management of toxicity.
* Signed informed consent from patients and/or their parents or legal guardians

Exclusion Criteria:

* Follicular lymphoma, MALT and nodular marginal zone are not included into this therapeutic study
* Patients with congenital immunodeficiency, chromosomal breakage syndrome, prior organ transplantation, previous malignancy of any type, or known positive HIV serology.
* Evidence of pregnancy or lactation period.
* There will be no exclusion criteria based on organ function.
* Past or current anti-cancer treatment except corticosteroids during less than one week.
* Tumor cell negative for CD20
* Prior exposure to rituximab.
* Severe active viral infection, especially hepatitis B.
* Hepatitis B carrier status history of HBV or positive serology.
* Participation in another investigational drug clinical trial.
* Patients who, for any reason, are not able to comply with the national legislation.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 482 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Event free survival | 24 months
  Minimum time to death from any cause, presence of viable cells in residue after [2nd (Rituximab-)CYVE], relapse, progressive disease, or second malignancy measured from randomization.

SECONDARY OUTCOMES:
Survival | 5 years
  Overall survival
Acute toxicity | 6 months
  Acute toxicity during treatment according to NCI-CTC V4
Long term toxicity | 5 years
  Long term toxicity, especially immune reconstitution, cardiac toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Véronique MINARD, MD, Study Chair — Institut Gustave Roussy, Villejuif, FRANCE; Thomas GROSS, MD, Study Chair — Children Oncology Group, USA
Locations (10):
- University Hospitals Leuven, Leuven, Belgium
- Children Oncology Group Operations centres, Monrovia, Canada
- The University of Hong Kong (Clinical Trials Centre), Hong Kong, China
- Institut de Cancérologie Gustave roussy, Villejuif, France
- 2nd Dept. of Pediatrics Semmelweis Univ., Budapest, Hungary
- Associazione Italiana di Ematologia ed Oncologia Pediatrica, Padua, Italy
- Emma Children's Hospital, Amsterdam, Netherlands
- Rectorat of Medical University, Wroclaw, Poland
- Sociedad Española de Hematología y Oncología Pediátricas, Valencia, Spain
- University of Birmingham, Birmingham, United Kingdom

REFERENCES:
- [Derived] Alexander S, Auperin A, Bomken S, Csoka M, Kazanowska B, Chiang AK, Andres M, Uyttebroeck A, Burke GAA, Zsiros J, Pillon M, Bollard CM, Mussolin L, Verdu-Amoros J, Neven B, Barkauskas DA, Wheatley K, Patte C, Gross TG, Minard-Colin V; Children's Oncology Group; European Intergroup for Childhood Non-Hodgkin's Lymphoma. Effect of rituximab on immune status in children with mature B-cell non-Hodgkin lymphoma: a prespecified secondary analysis of the Inter-B-NHL Ritux 2010 trial. Lancet Haematol. 2023 Jun;10(6):e445-e457. doi: 10.1016/S2352-3026(23)00062-5. Epub 2023 Apr 21. PMID 37094596
- [Derived] Lueza B, Auperin A, Rigaud C, Gross TG, Pillon M, Delgado RF, Uyttebroeck A, Amos Burke GA, Zsiros J, Csoka M, Simonin M, Patte C, Minard-Colin V, Bonastre J. Cost-effectiveness analysis alongside the inter-B-NHL ritux 2010 trial: rituximab in children and adolescents with B cell non-Hodgkin's lymphoma. Eur J Health Econ. 2024 Mar;25(2):307-317. doi: 10.1007/s10198-023-01581-y. Epub 2023 Apr 14. PMID 37058173
- [Derived] Minard-Colin V, Auperin A, Pillon M, Burke GAA, Barkauskas DA, Wheatley K, Delgado RF, Alexander S, Uyttebroeck A, Bollard CM, Zsiros J, Csoka M, Kazanowska B, Chiang AK, Miles RR, Wotherspoon A, Adamson PC, Vassal G, Patte C, Gross TG; European Intergroup for Childhood Non-Hodgkin Lymphoma; Children's Oncology Group. Rituximab for High-Risk, Mature B-Cell Non-Hodgkin's Lymphoma in Children. N Engl J Med. 2020 Jun 4;382(23):2207-2219. doi: 10.1056/NEJMoa1915315. PMID 32492302
- See also: Institute Gustave Roussy web site — http://www.igr.fr